CLINICAL TRIAL: NCT05966077
Title: Impact of Sending an Sms in the "Vigilans Lorraine" Monitoring System on the Rate of Telephone Responses of Subjects Contacted 3 Months After a Passage to the Suicidal Act
Brief Title: Impact of Sending an Sms on the Rate of Telephone Responses of Subjects Contacted 3 Months After the Suicidal Act
Acronym: EVAREST3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Psychothérapique de Nancy (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-A01404-39; RIPH-2022-02 (Other: Centre Psychothérapique de Nancy)
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-09

CONDITIONS: Suicide, Attempted
Keywords: suicide attempt prevention standby device
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: Randomized controlled trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS (Experimental): Sending an SMS 48 hours before the 3-month evaluation call planned as part of the VigilanS Lorraine system
  Interventions: Other: IMPACT OF SENDING AN SMS
- Without SMS (No Intervention): without Sending an SMS 48 hours before the 3-month evaluation call planned as part of the VigilanS Lorraine system

INTERVENTIONS:
Other: IMPACT OF SENDING AN SMS — Each subject of the experimental group will receive, in addition to the usual procedure of the VigilanS Lorraine device, an SMS 48 hours before the telephone call for evaluation at 3 months, warning him of this call.
  The time of this SMS has been set at 1:00 p.m. for all the people included in this group.
  At the end of this evaluation call, the caller will pass a satisfaction questionnaire to the subject in relation to the sending of the SMS
  Arms: SMS

SUMMARY:
The objective of this controlled, randomized, monocentric study is to compare the response rate of the call at 3 months of the groups with or without short message service (SMS) 48 hours before, for the subjects having benefited from the device "VigilanS Lorraine". The secondary objectives will be to appreciate the satisfaction of the subjects towards the sending of the SMS as well as to compare the delay of suicidal recidivism according to whether the subjects answered or not to the call of evaluation at 3 months of the passage to the act The main question it aims to answer is: What impact, on the rate of successful calls, could sending a text message 48 hours before the 3-month evaluation phone call have on subjects benefiting from the VigilanS device?

The participants will be divided into 2 groups:

* 1st group: SMS sent 48 hours before the 3-month evaluation call planned in the framework of the "VigilanS Lorraine" program.
* 2nd group (control): evaluation call at 3 months planned within the framework of the "VigilanS Lorraine" system, not preceded by an SMS 48 hours before.

The desired effect was an increase in the percentage of successful calls at 3 months, allowing for possible evaluations at 3 months in order to identify, evaluate and accompany subjects still in a suicidal crisis and thus avoid a recurrence of the act and thus a suicide.

ELIGIBILITY:
Inclusion Criteria:

* Having made a suicide attempt (first-time suicide or not)
* Hosted at the Central Hospital of Nancy
* Included in the "VigilanS Lorraine" monitoring system
* Not presenting criteria for non-inclusion in the "VigilanS Lorraine" system, namely:

  * Guardianship
  * Held
  * Dementia
  * Not speaking French
* Subject having received information relating to the progress of the EVAREST 3 study and having given their consent to participate
* Subject affiliated or entitled to a social security scheme

Exclusion Criteria:

* Subject without mobile phone
* Participation in another interventional study on the prevention of suicidal recidivism
* Subject under curatorship who was not assisted by his curator to give his consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of successful calls during the 3 month evaluation | 3 months
  . A call is considered unsuccessful after 3 call attempts at 3 different times over 3 consecutive working days.

SECONDARY OUTCOMES:
SMS delivery status: | 3 months
  issued/not issued
Satisfaction survey | 3 months
  subjective experience of the subject having benefited from the sending of the SMS in relation to the intervention, the delay between the sending of the SMS and the telephone call

CONTACTS AND LOCATIONS:
Overall Officials: Xavier SIPP, Mr., Principal Investigator — Centre Psychothérapique de Nancy

IPD SHARING:
Plan to Share IPD: No